CLINICAL TRIAL: NCT00817934
Title: Phase III of the AB Prep Safety and Efficacy in Colon Cleansing
Brief Title: Safe, Effective, and More Tolerable 16 Tablets Colon Prep
Acronym: ABP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Long Neck Medical Enterprises (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Semaan Abboud MD/ PI, Long Neck Medical Enterprises
Other Study IDs: ABBPREP1; AB1
Record Dates: First submitted 2009-01-05; First posted 2009-01-07 (Estimated); Last update posted 2009-01-07 (Estimated); Status verified 2009-01

CONDITIONS: Colon Cancer
Keywords: Efficacy; patient's tolerance; patient's safety
MeSH Terms: conditions — Colonic Neoplasms | interventions — Metoclopramide; Bisacodyl

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- PREVENTION AND TREATMENT: PATIENTS 50 YEARS AND OLDER REQUIRE SCREENING COLONOSCOPY. PATIENTS WITH FAMILY HISTORY OF COLON CANCER WILL REQUIRE IT BEFORE THE AGE OF 50.
  Interventions: Drug: AB PREP

INTERVENTIONS:
Drug: AB PREP — Potassium phosphate and Sodium Phosphate,(in the form of K-phos neutral 8 tablets.(Bisacodyl)6tablets. The third medication is (Metoclopramide).
  Other Names: Reglan, K-Phos neutral, and Dulcolax

SUMMARY:
The purpose of this study is determine if the AB Prep (a 16 tablets colon cleansing prep), is an effective, and safe colon cleansing prep in preparation for colonoscopy, and severe constipation.

DETAILED DESCRIPTION:
The available colon cleansing preps have issues with patient's tolerance( Abdominal pain, nausea, vomiting), and as recently noted by the FDA safety issues such a change in EKG, blood electrolytes requiring 72 hours to correct, and most recently PO4 nephropathy.

The AB Prep is a 16 tablets prep that has excellent patient's tolerance efficacy, with no change in blood electrolytes or EKG. ( PhaseI (20 patients) and Phase II (200 patients)

The protocol that was used is as follows:

(IND application # 75,704)

Protocol design for testing the safety and efficacy of the AB Prep:

The AB Prep is a combination of 2 Reglan tablets (10mg each), 6 Dulcolax tablets, and 8 K-Phos Neutral tablets. The combination is given in two steps, four hours apart; the day before the colonoscopy.

As before, the objective of this clinical trial is to examine the AB Prep first and foremost for safety, and second for efficacy of colon cleansing.

The proposed trial is for One-Arm Study of subjects undergoing elective and therapeutic colonoscopy.

Phase III: 400 patients, The selection will be random, the age probably ranging from 12 to 75 years old.

The patients will have a Pre, and post procedural EKG, comprehensive (Sodium, Potassium, Creatinine, BUN, Calcium, Magnesium, Phosphate, Glucose), and vital signs.

The patients with severe constipation (One bowel movement per week or more) will not be included in the study. (In our experience, those people required two days prep to achieve colon cleansing).

The SRSS statistical program will be used for data collection and analysis:

The end point of the study is colon cleansing, adequate enough to perform colonoscopy. The colon cleansing will be graded as follow:

1. Poor colon prep, unable to proceed with colonoscopy.
2. Able to do colonoscopy with, the colon cleansing labeled as:

A- Excellent, Totally cleansed B- Good, adequately cleansed, with need for irrigation.

In addition to efficacy, we would like to check for patient's satisfaction and compliance, (Most common complaints that the patients tend to voice with the present approved colon preps).

Patient's satisfaction data will be collected before the procedure and will be graded as follow:

1. Totally satisfied with the Prep, without any complaints
2. Satisfied, with the following complaints (Nausea, vomiting, abdominal pain/cramping)
3. Unsatisfied with the Prep (Reasons!!!)

Patient's compliance will be graded as follow:

1. Compliant
2. Non compliant(Reasons).

The prep instruction will be as follows REPARATION FOR COLONOSCOPY

FIVE DAYS before your procedure:

1. If you take COUMADIN or PLAVIX, we recommend that you stop these medications. You must contact your primary care physician or cardiologist for specific instructions. You may restart these medications again after the procedure unless otherwise instructed.
2. If you have DIABETES and take medication to control your blood sugar, contact your primary care physician or diabetes doctor for instructions about how to take your diabetes medication while preparing for this procedure.
3. Stop taking iron or multivitamins that contain iron.
4. Avoid the use of aspirin and aspirin-like medications such as ibuprofen, Advil and Aleve. These medicines may increase your risk of bleeding after polyp removal.
5. Start a low-roughage diet and do not eat corn or raw vegetables. You may re-start your usual diet after the procedure.

TWO DAYS before the procedure:

1. Take 2 tablets of Dulcolax at 8:00 PM.

ONE DAY before the procedure:

1. Begin a clear liquid diet at breakfast and continue this diet until 4 hours before your procedure. A clear liquid diet includes: water, tea, black coffee, clear broth, apple juice, white grape juice, Gatorade, soda, Jell-O. Do not eat or drink anything red, including red Jell-O. Do not drink milk. Do not use sugar-free drinks. All patients, including those with DIABETES, should be sure they get enough sugar during this time.
2. At 8:00 AM, take One Reglan(10mg) tablet, 2 Dulcolax tablets, and 4 tablets of K-PHOS NEUTRAL. Drink three glasses of water/juice SLOWLY over 1 hour. The laxative effect begins in about 2 hours. BE SURE TO DRINK AT LEAST 3 GLASSES OF WATER OR JUICE AFTER TAKING EACH DOSE OF THE prep.( Each Glass =350cc)
3. At 12:00 Noon, Take 2 Dulcolax tablets and 4 tablets of K-PHOS NEUTRAL, along with 3 glasses of water/Juice.(Each glass =350cc).

ON THE DAY of your procedure:

1. Take all of your usual medicines and 1 tablet of Reglan (10mg). Do Not Take Coumadin, Plavix, or Aspirin. If you take INSULIN, take 1/2 your usual dose.
2. If you have a medical condition requiring antibiotics before or after procedures, we will determine whether they are needed for your colonoscopy.
3. STOP CLEAR LIQUIDS 4 HOURS BEFORE YOUR PROCEDURE (except for small amount of water with medications). DO NOT EAT OR DRINK ANYTHING UNTIL AFTER YOUR PROCEDURE.
4. Wear loose-fitting, comfortable clothes.
5. Read the consent form. You will be asked to sign the form before your procedure.

Please bring these things WITH YOU to your procedure:

1. A list of all of your medications, including the doses
2. Your identification or insurance card
3. The name and phone number of your escort.

AFTER your procedure:

1. You will be monitored in the Endoscopy Unit recovery area for 20-30 minutes.
2. You may have some abdominal bloating after the procedure. It should resolve within an hour.

4. You may eat your normal diet after the procedure.

5. You may return to work the day after the procedure.

HELPFUL HINTS FOR PATIENTS UNDERGOING COLONOSCOPY

1.Use moist wipes (baby wipes) instead of toilet paper.

ELIGIBILITY:
Inclusion Criteria:

* Any eligible patient for colonoscopy

Exclusion Criteria:

* Patients with renal failure

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any patient between the age of 12 and 75, who is eligible for colonoscopy.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-01 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
TOTAL COLON CLEANSING, TO BE ABLE TO PERFORM COLONOSCOPY | IMMEDIATE, DURING THE COLONOSCOPY

CONTACTS AND LOCATIONS:
Overall Officials: SEMAAN M ABBOUD, MD, Principal Investigator
Locations (1):
- Cedar Tree Surgical Center, Millsboro, Delaware, United States